CLINICAL TRIAL: NCT04077931
Title: Blood Oxygenation Response to Aerobic and Breathing Exercises in Pregnant Women
Brief Title: Blood Oxygenation and Exercises in Pregnant Women
Acronym: exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Hany Farid Eid Morsy Elsisi (Unknown); yasser anees (Unknown)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoU7
Record Dates: First submitted 2019-08-31; First posted 2019-09-04 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-01

CONDITIONS: Aerobic and Breathing Exercises in Pregnant Women
Keywords: Aerobic; Exercises; Blood Oxygenation; Pregnancy
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: To investigate the blood oxygenation response to aerobic and breathing exercises in pregnant women. Participants and methods: A total of forty pregnant women participated in the study who were at the beginning of 3rd trimester. Their ages ranged from 25 to 30 years and their body mass index (BMI) was less than 30 kg/m2. They were assigned into two groups (A) performed aerobic exercises in a form of walking for 20-30 min. on treadmill at 60-75% of the target heart rate (THR) of each women, 3 times per week in addition to deep breathing exercises in form of diaphragmatic and lateral costal breathing, group (B) who performed deep breathing exercises only in form of diaphragmatic and lateral costal breathing. The program continued for 3 months, 3 times per week. The oxygen saturation (SaO2) was measured twice time firstly, at the beginning of 3rd trimester of pregnancy then after 3 months that at 24, 36 gestation weeks.
Who Masked: Outcomes Assessor
Masking Description: The women were randomly assigned to the treatment group(A) (n=25) or the control group (B) (n=25) by an independent person who selected numbers from sealed envelopes that containing numbers chosen by a random number generator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercises (Experimental): She asked to start walking with the speed of the machine was adjusted at 0.8 km/hour, so her resting pulse rate increases, then we increased the speed by 0.2 km/hour gradually every 2 minute (to give a time for adjustment of heart rate) till reaching our target heart rate (not less than 60% and not more than 75% of target heart rate). So the intensity of exercises can be increase or decrease only by changing the speed of treadmill according to target heart rate [13]
  Interventions: Other: exercises
- Deep breathing exercises (Experimental): Technique of breathing exercises: Regular aerobic exercises in a form breathing exercises included duration of 30 min. at 40-70% VO2 max. performed 2-3 per week. Each woman practiced deep breathing exercises 30 min. in the of form (diaphragmatic breathing exercises, 15 min. and lateral costal breathing exercises 15 min.) 3 times per week for 12 weeks.
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — Walking on treadmill with fixed 0% grade inclination

SUMMARY:
To investigate the blood oxygenation response to aerobic and breathing exercises in pregnant women. Participants and methods: A total of forty pregnant women participated in the study who were at the beginning of 3rd trimester. Their ages ranged from 25 to 30 years and their body mass index (BMI) was less than 30 kg/m2. They were assigned into two groups (A) performed aerobic exercises in a form of walking for 20-30 min. on treadmill at 60-75% of the target heart rate (THR) of each women, 3 times per week in addition to deep breathing exercises in form of diaphragmatic and lateral costal breathing, group (B) who performed deep breathing exercises only in form of diaphragmatic and lateral costal breathing. The program continued for 3 months, 3 times per week. The oxygen saturation (SaO2) was measured twice time firstly, at the beginning of 3rd trimester of pregnancy then after 3 months that at 24, 36 gestation weeks.

DETAILED DESCRIPTION:
Forty volunteers pregnant women at the beginning of 3rd trimester participated in this study. They were selected randomly from the gynecological outpatient clinic, at Kasr El Eini Universal Hospital, their ages were ranged from 25 to 30 years and body mass index indices (BMI) were less than 30 kg/m2. All participants were pregnant woman at the beginning of the 3rd trimester 12 weeks. Exclusion criteria of the study were as follows: Participant who had pulmonary diseases, cardiovascular diseases and psychiatric disorders.

Participants were assigned randomly used sealed envelope into two groups (A&B) equally in number. Group (A): Consisted of twenty pregnant woman at the beginning of the 3rd trimester. They performed aerobic exercise training in the form of walking on treadmill for 20 min, 3 times per week for 12 weeks. Then performed deep breathing exercises in form of diaphragmatic and lateral costal breathing. Group (B): Consisted of twenty pregnant woman at the beginning of the 3rd trimester who performed deep breathing exercises only in form of diaphragmatic and lateral costal breathing.

Methods Before the start of the first session, each pregnant woman was informed about program of exercises and informed consent form was signed from each woman before participation in the study. This study was conducted at from January 2018 to September 2019.

1-Aerobic exercises for all participants in group A: Women performed aerobic exercises in a form of walking for 20 min on treadmill 3 times per week for 12 weeks.

Treadmill: (power 220-V., 50/60 Hz): its speed, inclination and timer are adjustable and it also provided with control plane to display the exercises parameters

Intensity of exercises: The intensity of exercises was calculated as 60-75% of her target heart rate (THR) [11] (Q'Sullivan and Schmitz, 1999) as follow:

THR= {60-75% (HR max - HR rest)} + HR rest.

Where:

HR rest: resting heart rate in beat minute. MRH (Maximum heart rate=220 - Age in years) [12]

ELIGIBILITY:
Inclusion Criteria:

* their ages were ranged from 25 to 30 years
* body mass index (BMI) were less than 30 kg/m2

Exclusion Criteria:

* Participant who had pulmonary diseases
* cardiovascular diseases
* psychiatric disorders

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Pulse oxymeter | 12 weeks.
  It was used to measure oxygen saturation (SaO2) on the right index of each individual. Each individual sit quietly for about 5 minutes before the measurement and sit silently during the measurement.

CONTACTS AND LOCATIONS:
Overall Officials: ghada eb elrefaye, professor, Principal Investigator — Faculty of Physical therapy, Cairo University, Egypt.
Locations (1):
- Faculty of physical therapy- Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
investigate the blood oxygenation response to aerobic and breathing exercises in pregnant women
Supporting Information: Study Protocol
Time Frame: 3 months
Access Criteria: 3 months